CLINICAL TRIAL: NCT00906542
Title: Predictors of Early Chest Infection in Acute Ischemic Stroke
Acronym: PRECAST
Status: Completed | Type: Observational
Sponsor: University of Rostock (Other)
Responsible Party: Prof. Dr. Uwe Walter, University of Rostock, Department of Neurology
Other Study IDs: PRECAST-01
Record Dates: First submitted 2009-05-20; First posted 2009-05-21 (Estimated); Last update posted 2010-02-19 (Estimated); Status verified 2010-02

CONDITIONS: Acute Ischemic Stroke; Pneumonia
Keywords: acute stroke; ischemic stroke; pneumonia; chest infection; brain lesion; lesion topology; dysphagia; sympathetic activation; immunosuppression
MeSH Terms: conditions — Ischemic Stroke; Pneumonia; Stroke; Deglutition Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Acute ischemic stroke patients: Acute ischemic stroke patients admitted to the neurological intensive care unit or stroke unit within 24 hours after stroke onset in whom ischemic brain lesion was clearly assessed on CT and/or MRI

SUMMARY:
Pneumonia is a frequent complication of acute stroke and is associated with increased mortality and long-term impairment in the affected subjects. In previous studies, a number of clinical (e.g., dysphagia, severe neurological impairment, mechanical ventilation), radiological (e.g., large infarctions in the territory of middle cerebral artery, insular infarction) and biochemical (e.g., increased serum levels of C-reactive protein, decreased levels of CD4+ T-lymphocytes) findings have been reported as risk factors of stroke-related chest infection. The present study (PRECAST) aims to identify a small set out of these previously described risk factors that can predict stroke-related pneumonia with high sensitivity and specificity.

ELIGIBILITY:
Inclusion Criteria:

* acute ischemic stroke
* admission to the neurological intensive care unit or stroke unit within 24 hours after stroke onset
* clearly assessed brain lesion location

Exclusion Criteria:

* previous large (non-lacunar) stroke
* chest infection present already on hospital admission
* mechanical ventilation already on day 1 or 2 after hospital admission
* treatment with immunosuppressive drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute ischemic stroke patients admitted to the neurological intensive care unit or stroke unit within 24 hours after stroke onset
Sampling Method: Probability Sample
Enrollment: 530 (Actual)
Dates: Start 2009-05; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
diagnosis of chest infection within 7 days after stroke | days 1-7 after stroke

CONTACTS AND LOCATIONS:
Overall Officials: Uwe Walter, MD, Study Chair — University of Rostock, Germany
Locations (1):
- University of Rostock, Department of Neurology, Rostock, Germany

REFERENCES:
- [Background] Prass K, Meisel C, Hoflich C, Braun J, Halle E, Wolf T, Ruscher K, Victorov IV, Priller J, Dirnagl U, Volk HD, Meisel A. Stroke-induced immunodeficiency promotes spontaneous bacterial infections and is mediated by sympathetic activation reversal by poststroke T helper cell type 1-like immunostimulation. J Exp Med. 2003 Sep 1;198(5):725-36. doi: 10.1084/jem.20021098. Epub 2003 Aug 25. PMID 12939340
- [Background] Chamorro A, Amaro S, Vargas M, Obach V, Cervera A, Torres F, Planas AM. Interleukin 10, monocytes and increased risk of early infection in ischaemic stroke. J Neurol Neurosurg Psychiatry. 2006 Nov;77(11):1279-81. doi: 10.1136/jnnp.2006.100800. PMID 17043295
- [Background] Chamorro A, Amaro S, Vargas M, Obach V, Cervera A, Gomez-Choco M, Torres F, Planas AM. Catecholamines, infection, and death in acute ischemic stroke. J Neurol Sci. 2007 Jan 15;252(1):29-35. doi: 10.1016/j.jns.2006.10.001. Epub 2006 Nov 28. PMID 17129587
- [Background] Walter U, Knoblich R, Steinhagen V, Donat M, Benecke R, Kloth A. Predictors of pneumonia in acute stroke patients admitted to a neurological intensive care unit. J Neurol. 2007 Oct;254(10):1323-9. doi: 10.1007/s00415-007-0520-0. Epub 2007 Mar 14. PMID 17361338
- [Background] Vogelgesang A, Grunwald U, Langner S, Jack R, Broker BM, Kessler C, Dressel A. Analysis of lymphocyte subsets in patients with stroke and their influence on infection after stroke. Stroke. 2008 Jan;39(1):237-41. doi: 10.1161/STROKEAHA.107.493635. Epub 2007 Nov 29. PMID 18048864
- [Background] Steinhagen V, Grossmann A, Benecke R, Walter U. Swallowing disturbance pattern relates to brain lesion location in acute stroke patients. Stroke. 2009 May;40(5):1903-6. doi: 10.1161/STROKEAHA.108.535468. Epub 2009 Mar 12. PMID 19286597